CLINICAL TRIAL: NCT01024400
Title: Etude de Phase II évaluant l'immunogénicité et la tolérance d'un Vaccin inactivé Non adjuvanté Contre la Grippe A(H1N1)v Chez la Femme Enceinte
Brief Title: Immunogenicity and Safety of an Inactivated Non-adjuvanted A(H1N1)v Influenza Vaccine in Pregnant Women
Acronym: PREFLUVAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C09-33; 2009-016660-36 (EudraCT Number)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2011-03

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Pregnancy
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccine (Experimental)
  Interventions: Biological: Non-adjuvanted A(H1N1)v influenza vaccine

INTERVENTIONS:
Biological: Non-adjuvanted A(H1N1)v influenza vaccine — 15 mcg HA/0.5 ml

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of an inactivated, non adjuvanted A(H1N1)v influenza vaccine in 120 pregnant women.

Study procedures will include 2 doses of vaccine, blood samples, cord blood samples at delivery and recording temperature and vaccine side effects in a memory aid for 7 days following each vaccination. Participants will be involved in study related procedures about 3 at 5 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 45 years
* Pregnancy between 22 and 32 weeks of gestation
* Provides written informed consent
* Covered by French Social Security

Exclusion Criteria:

* Allergy to eggs or other components in the vaccine
* History of severe reactions following previous influenza vaccines
* H1N1 influenza (virologically documented) during the last 6 months
* Febrile episode within one week prior to vaccination
* Known HIV, HBV, HCV infection
* Multiple sclerosis
* History of Guillain-Barré syndrome
* Organ transplant recipient
* Neoplastic disease in the past 3 years
* Other vaccine within 3 weeks prior to study entry or planned within the month following the last injection
* Systemic corticosteroids,immunotherapy,chemotherapy
* Anticoagulant treatment
* Immunoglobulin or blood transfusion within the 3 months prior to enrollment in this study
* History of cardiac disease
* Chronic liver disease
* Diabetes before pregnancy
* History of premature delivery
* History of eclampsia
* Fetal morphologic abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: proportion of subjects achieving a serum HAI antibody titer of greater than or equal to 1:40, proportion of subjects with 4-fold or greater HAI antibody titer increases against H1N1 2009 virus following H1N1 vaccine. | Day 21

SECONDARY OUTCOMES:
Safety: occurence of local and systemic adverse events | Throughout the course of the study
Immunogenicity: proportion of subjects achieving a serum HAI antibody titer of greater than or equal to 1:40, proportion of subjects with 4-fold or greater HAI antibody titer increases against H1N1 2009 virus following H1N1 vaccine. | Day 42 and at delivery
Safety:occurence of vaccine-associated serious adverse events | Throughout the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, Principal Investigator — Groupe hospitalier Cochin Saint Vincent de Paul; Vassilis Tsatsaris, MD, Principal Investigator — Groupe hospitalier Cochin Saint Vincent de Paul
Locations (5):
- France (5):
  - CHU de Besançon-Hôpital Saint-Jacques, Besançon
  - Hôpital Antoine Béclère, Clamart
  - Groupe hospitalier Cochin Saint Vincent de Paul, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Sud de Rennes, Rennes

REFERENCES:
- [Result] Tsatsaris V, Capitant C, Schmitz T, Chazallon C, Bulifon S, Riethmuller D, Picone O, Poulain P, Lewin F, Laine F, Jacqz-Aigrain E, Aboulker JP, Launay O; Inserm C09-33 PREFLUVAC (Immunogenicity and Safety of an Inactivated Nonadjuvanted A[H1N1v] Influenza Vaccine in Pregnant Women) Study Group. Maternal immune response and neonatal seroprotection from a single dose of a monovalent nonadjuvanted 2009 influenza A(H1N1) vaccine: a single-group trial. Ann Intern Med. 2011 Dec 6;155(11):733-41. doi: 10.7326/0003-4819-155-11-201112060-00005. PMID 22147712